CLINICAL TRIAL: NCT02593903
Title: Prophylactic Antibiotics Following Distal/Mid-shaft Hypospadias Repair: Are They Necessary?
Brief Title: Antibiotic Use Following Distal and Mid-shaft Hypospadias Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Children's Hospital and Health System Foundation, Wisconsin (Other)
Responsible Party: Principal Investigator, Travis Groth, Assistant Professor, MD, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHW 13/140
Record Dates: First submitted 2015-10-30; First posted 2015-11-02 (Estimated); Results first posted 2018-11-05 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Hypospadias
Keywords: Antibiotic Prophylaxis
MeSH Terms: conditions — Hypospadias | interventions — Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antibiotics Group (Experimental): Patients randomized to this arm will receive prophylactic oral antibiotics following the surgery and catheter placement (Septra, 3 mg/kg/dose once daily), and will continue the medication for until the day before catheter removal 4-8 days post-operation.
  Interventions: Drug: Septra
- No Antibiotics Group (No Intervention): Patients randomized to this arm will receive regular clinical care without prophylactic antibiotics, including catheter placement/removal.

INTERVENTIONS:
Drug: Septra
  Other Names: Bactrim; Sulfamethoxazole/trimethoprim
  Arms: Antibiotics Group

SUMMARY:
The purpose of this study is to evaluate the efficacy of prophylactic antibiotics following distal or mid-shaft hypospadias repair in influencing the rate of postoperative urinary tract infection and complications.

DETAILED DESCRIPTION:
The rationale for using prophylactic antibiotics after hypospadias surgery is to decrease the occurrence of urinary tract infections (UTIs) and complications. However, even though prophylactic antibiotics are used by some pediatric urologists, to date there has been no evidence supporting the role of prophylactic antibiotics in decreasing UTIs or complications. This is a prospective, randomized trial involving children undergoing distal or mid-shaft hypospadias repair. Subjects randomized into a group taking prophylactic dosages of antibiotics and a group not receiving post-operative antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* all children between ages 6 months to 2 years under going distal or mid shaft hypospadias repair
* children of parents who give informed consent
* English speaking
* participant must be available for follow-up 3 and 12 months post-surgery

Exclusion Criteria:

* all proximal hypospadias and redo hypospadias repairs
* children who are allergic to sulfa medications
* patients who have UTI at time of surgery (proven by culture)

Ages: 6 Months to 2 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 67 (Actual)
Dates: Start 2014-03-04 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Travis W Groth, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Background] Meir DB, Livne PM. Is prophylactic antimicrobial treatment necessary after hypospadias repair? J Urol. 2004 Jun;171(6 Pt 2):2621-2. doi: 10.1097/01.ju.0000124007.55430.d3. PMID 15118434
- [Derived] Roth EB, Kryger JV, Durkee CT, Lingongo MA, Swedler RM, Groth TW. Antibiotic Prophylaxis with Trimethoprim-Sulfamethoxazole versus No Treatment after Mid-to-Distal Hypospadias Repair: A Prospective, Randomized Study. Adv Urol. 2018 Mar 26;2018:7031906. doi: 10.1155/2018/7031906. eCollection 2018. PMID 29780414

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Antibiotics Group | No Antibiotics Group
Started | 35 | 32
Completed | 35 | 31
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Antibiotics Group | No Antibiotics Group | Total
Number analyzed (Participants) | 35 | 32 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 35 | 32 | 67
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 35 | 32 | 67
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Urinary Tract Infection
Description: Urinary tract infection (UTI) will be diagnosed based on urine culture positive at 50,000CFUs per mL with one or both of the following: fever >38 Celsius, or significant fussiness and irritability with voiding per parent report. Asymptomatic bacteriuria is known and expected in this population; therefore culture positive results alone will not be sufficient to meet the definition of UTI.
Time Frame: 4-8 days post-operation
Population: Out of the consented and randomized participants these were the patients that we were able to obtain a post Op Urine sample
Measure: Count of Participants; unit: Participants
Arm/Group | Antibiotics Group | No Antibiotics Group
Number analyzed (Participants) | 30 | 22
Participants
  Post Op Urine Sample obtained | 30 | 22
  clinical UTI | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Antibiotics Group | No Antibiotics Group
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/32
Other Adverse Events (participants affected / at risk) | 0/35 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-12-16): https://cdn.clinicaltrials.gov/large-docs/03/NCT02593903/Prot_SAP_000.pdf